CLINICAL TRIAL: NCT01158677
Title: Short Term Outcome After Meniscectomy
Status: Completed | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: 2010/117
Record Dates: First submitted 2010-07-07; First posted 2010-07-08 (Estimated); Last update posted 2022-12-14 (Actual); Status verified 2022-12

CONDITIONS: Meniscectomy
Keywords: meniscectomy
MeSH Terms: interventions — Meniscectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Meniscectomy — patients undergoing meniscectomy will be asked to complete the KOOS-scale,Vas-scale, Tegner questionnaire, SF-36 questionnaire pre-operatively and at 3, 6 and 12 months post-operatively

SUMMARY:
Short term outcome after meniscectomy: a meniscectomy is a very frequent performed orthopedically procedure. The short term outcome is favourable, but some patients keep having residual lesions after surgery.

This prospective study examens the clinical outcome after meniscectomy using questionnaires (KOOS, VAS, SF-36, Tegner) (before the surgery, 3, 6 & 12 months postoperative.) The investigators will also record the further treatment options for the people at risk.

ELIGIBILITY:
Inclusion criteria:

* all the meniscectomy patients (male & female, all ages)

Exclusion Criteria:None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all the meniscectomy patients (male & female, all ages)
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2010-07 (Actual); Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
The clinical outcome (residual lesions) after a meniscectomy | 12 months post-operative
  KOOS-scale, Vas-scale, Tegner questionnaire, SF-36 questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Peter Verdonk, MD, Principal Investigator — University Hospital Ghent, Belgium
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- See also: website of University Hospital Ghent, Belgium — http://www.uzgent.be